CLINICAL TRIAL: NCT01956890
Title: Integrative Diagnosis of 18F-FLT Positron Emission Tomography and Magnetic Resonance Imaging to Evaluate the Suspicious Findings on Mammography and Breast Ultrasound: a Pilot Study
Brief Title: 18F-FLT Positron Emission Tomography and Magnetic Resonance Imaging of the Breast
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 201102011MB
Record Dates: First submitted 2013-09-24; First posted 2013-10-08 (Estimated); Last update posted 2013-10-16 (Estimated); Status verified 2013-10

CONDITIONS: Breast Cancer
Keywords: Breast neoplasms; PET; MRI
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- diagnostic accuracy (Other): diagnostic accuracy of PET and MRI for breast cancer diagnosis.
  Interventions: Drug: PET

INTERVENTIONS:
Drug: PET — 18F-FLT PET and MRI of the breast
  Other Names: 3'-deoxy-3'-[18F]fluorothymidine PET

SUMMARY:
This prospective study is aimed to evaluate the diagnostic effectiveness of 18F-FLT PET in differentiating benign nature from malignancy for lesions with suspicious or ambiguous findings on mammography or ultrasound; to determine whether 18F-FLT PET or MRI can increase the specificity in breast lesion diagnosis and thus reduce the unnecessary biopsy, and which (18F-FLT PET or MRI) reveals the higher diagnostic performance.

DETAILED DESCRIPTION:
It has been reported that PET (Positron Emission Tomography) scan is also useful in diagnosing breast cancer. 18F-fluorodeoxyglucose (18F-FDG), which based on glucose metabolism for the determination of malignancy, is the most popular PET tracer at present. However, 18F-FDG is not tumor specific. Benign inflammatory lesions may also demonstrate increase in 18F-FDG uptake. On the other hand, low grade malignancy may have low 18F-FDG concentration. Recently, 18F-3'-fluoro-3'-deoxy-L-thymidine (18F-FLT), a radiolabelled analog of thymidine, has been used in imaging cell proliferation and monitoring of treatment effects for breast cancer patients. 18F-FLT is believed to be more specific than 18F-FDG for breast cancer diagnosis and may provide the underlined physiological and molecular manifestations of breast lesions in addition to anatomical manifestations from mammography, ultrasound or MRI. Yet, its potential role in differentiation of ambiguous or suspicious lesions found on conventional imaging, such like mammography or ultrasound, has not been reported. We have had an ongoing preliminary study regarding breast lesion diagnosis using 18F-FLT PET, with an overall sensitivity 100% and specificity 92.7% in this dataset (from 2010 August to 2010 December, 19 lesions from 8 women with correlation with biopsy and clinical outcome).

On the other hand, the molecular subtypes of breast cancer, including ER (Estrogen receptor), PR (Progesterone receptor), HER2 (Human epidermal growth factor receptor 2) are associated with treatment planning and prediction of clinical outcome of breast cancer. There have been documented reports regarding the relation of mammography, DCE MRI, 18F-FDG PET to ER, PR, HER2 status of breast cancers. But the association of proton MRS, DWI and 18F-FLT PET with ER, PR, HER2 status was seldom reported.

ELIGIBILITY:
Inclusion Criteria:

* 1) Women aged between 20 to 80 years 2) women who have localized findings on mammography and / or ultrasound and will receive biopsy 3) The lesions on the conventional imaging measure >=1cm 4) WBC count >=3000/L, or platelet>=75,000/L 5) Liver function, AST or ALT <78 U/L 6) Renal function, Creatinine <2.0 mg/dl., and estimated GFR(eGFR)>60ml/min/1.73m2.

Exclusion Criteria:

* 1) Pregnant women or who are planning to be pregnant, or who are lactating. (Eligible women who are premenopausal with reproductive potential should receive urine pregnancy test before the MRI and PET. Women with a positive pregnancy test should be excluded from the study.) 2) Known cancers in other organs. 3) Women who are not able to cooperate with the PET/CT examination, or MRI examination.

  4) Women≦19 years old. 5) Past history of severe anaphylactoid reaction to MRI-contrast agent or 18F-FLT.

  6) History of mechanical valve replacement, recent coronary artery stent placement, with pacemaker, aneurysmal clip, metallic endotracheal tube, or other procedures with metallic device application.

  7) eGFR≦60ml/min/1.73m2. 8) History of acute renal failure, or renal dialysis.

Ages: 20 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2011-06; Primary Completion 2015-12 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
diagnostic accuracy of 18F-FLT PET and MRI | 5 years
  to measure diagnostic accuracy (sensitivity, specificity) of 18F-FLT PET and MRI for localized breast findings seen on mammography and breast ultrasound.

CONTACTS AND LOCATIONS:
Overall Officials: Jane Wang, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan, Taiwan